CLINICAL TRIAL: NCT04491513
Title: Detection of Proximal Coronary Artery Disease in the Work-up for Transcatheter Aortic Valve Implantation Using CTA (From the DEPICT CTA Database)
Acronym: DEPICT CTA
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, J.P.S Henriques, Prof, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: Amsterdam UMC
Record Dates: First submitted 2020-07-26; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Computed Tomography Angiography; Coronary Artery Disease; Coronary Angriography; Aortic Valve Disease
Keywords: Computed tomography angiography; coronary angriography; Aortic Valve Disease; Transcatheter aortic valve implantation
MeSH Terms: conditions — Coronary Artery Disease; Aortic Valve Disease | interventions — Computed Tomography Angiography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Overall cohort: Pateints that underwent both CTA and CAG in the work-up for TAVI
  Interventions: Diagnostic Test: Computed tomography angiography

INTERVENTIONS:
Diagnostic Test: Computed tomography angiography — Computed tomography angiography for the detection of proximal coronary lesions in patients in the work-up for TAVI

SUMMARY:
Background: Computed tomography angiography (CTA) is already used in the work-up for transcatheter aortic valve implantation (TAVI) and could partially replace invasive coronary angiography (CAG) to rule out proximal coronary lesions.

Objectives: To assess the diagnostic accuracy and yield of pre-TAVI CTA to detect coronary lesions (≥50% DS and ≥70% DS) in the proximal coronary segments on a per-patient and a per-segment level.

Methods: The DEPICT CTA database consists of individual patient data of four studies that analysed the diagnostic accuracy of pre-TAVI CTA to detect coronary lesions. For this analysis, diagnostic accuracy was assessed in the left main and the three proximal coronary segments.

DETAILED DESCRIPTION:
Methods Objectives To assess the diagnostic accuracy and yield of pre-TAVI CTA to detect coronary lesions (≥50% DS and ≥70% DS) in the proximal coronary segments on a per-patient and a per-segment level. The secondary objective was to perform a subgroup analysis of the individual included studies and to assess the influence of atrial fibrillation and heart rate on the diagnostic accuracy.

Literature search and study selection Studies were selected from our previous systematic review and meta-analysis on the diagnostic accuracy of CTA for the detection of significant CAD in TAVI work-up [4]. These studies were supplemented with studies that were retrieved by an updated literature search in OVID MEDLINE (including Epub Ahead of Print, In-Process & Other Non-Indexed Citations) and OVID EMBASE from January 1, 1946 to October 01, 2019. Studies were excluded if they were not reporting original data of patients who received both pre-procedural multi-detector computed tomography (MDCT) and CAG for the evaluation of CAD in the work-up of TAVI. The authors of 8 studies were approached to jointly perform a meta-analysis of individual patient data. The authors of 4 studies could accommodate the data for a per segment analysis [5-8]. The methodological quality of the included studies was assessed using the modified Quality Assessment of Studies of Diagnostic Accuracy Included in Systematic Reviews-2 criteria (QUADAS-2) [9].

Data collection The data sets included patient characteristics regarding age, sex, body mass index (BMI) and the heart rate during CT-scan. Information about co-morbidities included the presence of diabetes mellitus, atrial fibrillation, hypercholesterolemia, peripheral atrial disease, hypertension, a history of smoking, presence of CAD and a history of PCI or coronary artery bypass grafting. Technical CT scanner information included scanner type, number of detector rows, number of slices, detector width, CT scanner rotation time, scan protocol and settings (tube voltage and tube current), contrast agent type and volume, dose length product, and nitroglycerine use.

The coronary segments were categorized in three categories: lesions <50% DS, lesion ≥50-70% DS or lesions ≥70% DS), according to the 18-segment coronary model of the Society of Cardiovascular Computed Tomography or the American Heart Association modified 15-segment model [10,11]. All studies used a cut-off of ≥50% diameter stenosis to determine the presence of obstructive CAD. Three out of four studies also used a cut-off value of ≥70% DS [5,7,8], which were used for an additional analysis of the diagnostic accuracy to detect ≥70% DS proximal obstructive coronary lesions. If a segment had poor image quality or severe motion artefacts, it was labelled as non-diagnostic.

Statistical analysis Data analysis was performed using the statistical software R version 3.5.1 (R Foundation for Statistical Computing, Vienna, Austria). Continuous variables were presented as means with standard deviations (SD). The distribution of continuous variables was tested with the Shapiro-Wilk test. Categorical variables were presented as frequencies and percentages. The prevalence of proximal lesions of ≥50% DS and of ≥70% DS was computed from the measurements with invasive CAG, because revascularization with PCI is only considered in case of a proximal ≥70% DS lesion.(ref ESC guideline) Diagnostic accuracy of pre-TAVI CTA, as compared to pre-TAVI CAG, was defined as the sensitivity, specificity, positive - (PPV) and negative predictive value (NPV) and was derived from the number of true positives (TP), true negatives (TN), false positives (TP) and false negatives (FN). The analysis of the primary endpoint was performed on a per-patient and per-segment level. Diagnostic accuracy was computed for CTA to detect obstructive proximal coronary lesions of more than 50% DS and also of ≥70% DS lesions in a subgroup of patients were the data was available. All non-diagnostic segments were considered as abnormal tests and were labelled as if there was a lesion. For the per-patient analysis of diagnostic accuracy, patients were regarded as having proximal obstructive lesions if there was a minimum of one non-diagnostic segment. Diagnostic yield was defined as the number of patients that would not need an invasive CAG if pre-TAVI CTA was used as a gatekeeper to rule out obstructive proximal lesions and was derived from the sum of the negatives (TN + FN). For the subgroup analysis, we analysed the diagnostic accuracy in the individual included studies and assessed the diagnostic accuracy in the subgroups with atrial fibrillation and a heart rate <70 and ≥70 b/min. The diagnostic accuracy in the individual studies and the subgroups was assessed on a per-patient level for lesions ≥50% DS.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the work-up for TAVI

Exclusion Criteria:

* inability to undergo CTA

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients in the work-up for TAVI
Sampling Method: Probability Sample
Enrollment: 1060 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy and yield of pre-TAVI CTA to detect coronary lesions (≥50% DS and ≥70% DS) in the proximal coronary segments on a per-patient and a per-segment level. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data will be made available during or after publication of initial outcome paper
Supporting Information: Study Protocol, SAP
Time Frame: data will be made available upon publication

REFERENCES:
- [Background] Andreini D, Pontone G, Mushtaq S, Bartorelli AL, Ballerini G, Bertella E, Segurini C, Conte E, Annoni A, Baggiano A, Formenti A, Fusini L, Tamborini G, Alamanni F, Fiorentini C, Pepi M. Diagnostic accuracy of multidetector computed tomography coronary angiography in 325 consecutive patients referred for transcatheter aortic valve replacement. Am Heart J. 2014 Sep;168(3):332-9. doi: 10.1016/j.ahj.2014.04.022. Epub 2014 Jun 9. PMID 25173545
- [Background] Opolski MP, Kim WK, Liebetrau C, Walther C, Blumenstein J, Gaede L, Kempfert J, Van Linden A, Walther T, Hamm CW, Mollmann H. Diagnostic accuracy of computed tomography angiography for the detection of coronary artery disease in patients referred for transcatheter aortic valve implantation. Clin Res Cardiol. 2015 Jun;104(6):471-80. doi: 10.1007/s00392-014-0806-z. Epub 2015 Jan 6. PMID 25559245
- [Background] Hamdan A, Wellnhofer E, Konen E, Kelle S, Goitein O, Andrada B, Raanani E, Segev A, Barbash I, Klempfner R, Goldenberg I, Guetta V. Coronary CT angiography for the detection of coronary artery stenosis in patients referred for transcatheter aortic valve replacement. J Cardiovasc Comput Tomogr. 2015 Jan-Feb;9(1):31-41. doi: 10.1016/j.jcct.2014.11.008. Epub 2014 Dec 3. PMID 25576406
- [Background] Rossi A, De Cecco CN, Kennon SRO, Zou L, Meinel FG, Toscano W, Segreto S, Achenbach S, Hausleiter J, Schoepf UJ, Pugliese F. CT angiography to evaluate coronary artery disease and revascularization requirement before trans-catheter aortic valve replacement. J Cardiovasc Comput Tomogr. 2017 Sep-Oct;11(5):338-346. doi: 10.1016/j.jcct.2017.06.001. Epub 2017 Jun 22. PMID 28662835